CLINICAL TRIAL: NCT05675670
Title: Artificial Intelligence-enable Electrocardiogram for Diagnosis and Outcome in Hyperthyroidism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2022001
Record Dates: First submitted 2022-12-26; First posted 2023-01-09 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will have access to the screening tool
  Interventions: Other: AI-enabled ECG-based Screening Tool
- Control (No Intervention): Patients randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool — Primary care clinicians in the intervention group had access to the report, which displayed whether the AI-ECG result was positive or negative. The system will send a message to corresponding physicians if positive finding.
  Arms: Intervention

SUMMARY:
hyperthyroidism

ELIGIBILITY:
Inclusion Criteria:

* Patients in outpatient department.
* Patients recieved at least 1 ECG examination.
* Patients without TSH test before ECG examination or patients with subclinical hyperthyroidism without anti-thyroid drug usage.

Exclusion Criteria:

* The patients recieved ECG at the period of inactive AI-ECG system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
New-onset hyperthyroidism | Within 30 days
  A TSH of <0.25 IU/L
New-onset anti-throid drug treatment | Within 60 days
  New anti-throid drug treatment for patients with subclinical hyperthyroidism

SECONDARY OUTCOMES:
All-cause mortality | Within 1 year.
  All-cause mortality
Cardiac event | Within 1 year.
  Heart failure, arrhythmia, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No